CLINICAL TRIAL: NCT03213145
Title: A Non-Randomized, Open-Label, Two-Part, Drug-Drug Interaction Study to Evaluate the Effects of Itraconazole and Rifampin on the Pharmacokinetics and Safety of EDP-305 in Healthy Volunteers
Brief Title: Drug-drug Interaction Study Between EDP-305, Intraconazole and Rifampin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EDP 305-005
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-07

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
Keywords: drug-drug interaction
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Rifampin

STUDY DESIGN:
Intervention Model Description: 2-Part Single Group study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Experimental)
  Interventions: Drug: intraconazole; Drug: EDP 305
- Part 2 (Experimental)
  Interventions: Drug: Rifampin; Drug: EDP 305

INTERVENTIONS:
Drug: intraconazole — Subjects will receive itraconazole once daily from Day 5 through Day18
  Arms: Part 1
Drug: Rifampin — Subjects will receive rifampin once daily from Day 5 through Day 16
  Arms: Part 2
Drug: EDP 305 — Subjects will receive EDP 305 once daily on Day 1 and Day 14

SUMMARY:
This is a non-randomized, 2-part, open-label, drug-drug interaction (DDI) study to evaluate the effect of concomitant administration of itraconazole or rifampin on the pharmacokinetics and safety of EDP-305 in healthy human volunteers.

ELIGIBILITY:
Inclusion Criteria:

* An informed consent document signed and dated by the subject.
* Healthy male and female subjects of any ethnic origin between the ages of 18 and 55 years, inclusive.
* Female subjects must be of non-childbearing potential.

Exclusion Criteria:

* Clinically relevant evidence or history of illness or disease.
* Pregnant or nursing females.
* History of febrile illness within 7 days prior to the first dose of study drug or subjects with evidence of active infection.
* A positive urine drug screen at screening or Day -1.
* Current tobacco smokers or use of tobacco within 3 months prior to screening.
* Any condition possibly affecting drug absorption (e.g., gastrectomy, cholecystectomy).
* History of regular alcohol consumption.
* Participation in a clinical trial within 30 days prior to the first dose of study drug.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2017-08-10 (Actual); Study Completion 2017-09-07 (Actual)

PRIMARY OUTCOMES:
Cmax of EDP-305 with and without coadministration with itraconazole | Up to 19 days
AUC of EDP-305 with and without coadministration with itraconazole | Up to 19 days
Cmax of EDP-305 with and without coadministration with rifampin | Up to 17 days
AUC of EDP-305 with and without coadministration with rifampin | Up to 17 days

SECONDARY OUTCOMES:
Safety measured by adverse events, physical exams, vital signs, 12-lead electrocardiograms (ECGs) and clinical lab results (including chemistry, hematology, and urinalysis). | Up to 19 days

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Inc, Study Director — Enanta Pharmaceuticals, Ind
Locations (1):
- Pharmaceutical Research Associates, Inc.,, Lenexa, Kansas, United States